CLINICAL TRIAL: NCT05971121
Title: Comparing Ciprofol and Propofol for Sedation in Hypotensive ICU Patients: a Single Center Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-525
Record Dates: First submitted 2023-05-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Ciprofol; Propofol; Sedation; Low Blood Pressure; Norepinephrine
MeSH Terms: conditions — Hypotension | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ciprofol group: Hypotensive ICU patient sedated with ciprofol
  Interventions: Drug: ciprofol
- propofol group: Hypotensive ICU patient sedated with propofol

INTERVENTIONS:
Drug: ciprofol — Ciprofol were used for sedation in ICU hypotensive patients
  Groups: ciprofol group

SUMMARY:
This study was a single-center, prospective, 2-year observational cohort study. The study subjects were ICU patients requiring vasopressor drugs and requiring sedation. According to the use of ciprofol or propofol in the treatment plan (determined by the doctor in charge according to the condition of the subjects), they were divided into groups: ciprofol group and propofol group. A total of 456 subjects were planned to be enrolled, including 304 subjects in the cyclopofol group and 152 subjects in the propofol group. The data of this study were obtained by extracting the routine clinical diagnosis and treatment records of the enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* It needs to be treated with vasopressors to maintain mean arterial pressure ≥65 mmHg;
* Sedative medication required for comfort, safety, and to facilitate life support measures;
* Obtain the informed consent of the human subjects or their legal representatives.

Exclusion Criteria:

* Pregnant patient;
* Patients with proven acute severe intracranial or spinal neurological disease due to vascular, intracranial dilatation, or injury;
* History of allergy to cyclopofol, propofol, eggs, or soy products;
* History of long-term use of benzodiazepines or opioids;
* Sedative drugs other than propofol or cyclopofol were used at enrollment, or propofol and cyclopofol were used alternately within 24 hours;
* The researchers judged that they are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Department of Critical Care Medicine, Nanfang Hospital, Southern Medical University, patients needing vasopressor drugs to maintain blood pressure while requiring sedation
Sampling Method: Probability Sample
Enrollment: 456 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients meeting the RASS sedation | within 24 hours
  Professionally trained researchers perform RASS scores on patients at specific time points

SECONDARY OUTCOMES:
Dosage of propofol or ciprofol during sedation (total dose/time of use) | up to 24 hours
  Responsible researchers consult the patient's medical record after completing treatment to obtain the dosage and duration of medication
Dosage of norepinephrine during sedation (total dose/time of use) | up to 24 hours
  Responsible researchers consult the patient's medical record after completing treatment to obtain the dosage and duration of medication
Duration of mechanical ventilation | From endotracheal intubation to withdrawal from mechanical ventilation,up to 28 days
  Responsible researchers obtain information by viewing electronic medical records
Incidence of adverse events | up to 3 days
  The occurrence of adverse events during the hospital period will be recorded in the medical record by the clinician or nurse, and the researcher will obtain the occurrence of adverse events (event type, time, treatment, results, etc.) through the medical record
length of ICU stay | up to 28 days
  Researchers obtain it through the hospital electronic system
The mortality rate | up to 28 days
  Researchers obtain it through the hospital electronic system.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern medical university Nanfang hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided